NCT04031105 ECS Kranz: Priming TBS 20220329

## CONSENT TO PARTICIPATE IN RESEARCH

Title of Research Project

## PROBING HOMEOSTATIC PLASTICITY WITH PRIMING THETA-BURST STIMULATION OF THE DORSOLATERAL PREFRONTAL CORTEX

| Iher | beby consent to participant in the captioned research |
|---|---|
| conducted by | |
| | from this research may be used in future research and y will be retained, i.e. my personal details will not be |
| • | information sheet has been fully explained. I understand |
| the benefit and risks involved. My partici | pation in the project is voluntary. |
| I acknowledge that I have the right to que<br>time without penalty of any kind. | estion any part of the procedure and can withdraw at any |
| Name of participant | |
| Signature of participant | |
| Name of researcher | |
| Signature of researcher | |
| Date | |